CLINICAL TRIAL: NCT05194436
Title: A Pilot Study to Assess Aevice Medical Device for Detection of Wheeze in Pediatric Subjects and Use for Remote Auscultation
Brief Title: Wheeze Detection Using Aevice Medical Device
Status: Completed | Type: Observational
Sponsor: Aevice Health Pte. Ltd. (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: AE_MD_001
Record Dates: First submitted 2021-12-17; First posted 2022-01-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Subject Presenting Wheeze; COPD; Asthma
Keywords: Wheeze; Auscultation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: AeviceMD — The AeviceMD will be placed on the patient to detect wheeze and perform auscultation.
  Other Names: AeviceMD Monitoring System

SUMMARY:
The primary objective of this study is to determine if Aevice Medical Device can detect wheeze as accurately as a physician through auscultation. The secondary objective is to investigate if Aevice Medical Device can be used for remote auscultation of the lung.

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing and parents/guardians are able to give informed consent for participation in the study.
* Male or Female, aged 3 -18 years.
* Presenting with wheeze.
* Able (in the Investigators opinion) and willing to comply with all study requirements

Exclusion Criteria:

* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the subjects at risk because of participation in the study, or may influence the result of the study, or the subject's ability to participate in the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study will include 35 patients who are admitted for exacerbations of chronic airway disease (i.e. Asthma)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Wheeze is detected by physician and AeviceMD | 60 Seconds
  Primary end point of wheeze will be captured in a binary fashion (i.e. PRESENT or NOT PRESENT) on the CRF by the physician during manual auscultation. AeviceMD will perform wheeze analysis on each 5 sec of recording

SECONDARY OUTCOMES:
Respiratory sounds are detected and identified by onsite physician and offsite (remote) physician | 150 Seconds
  Secondary end point of normal, adventitious and lack of breath sounds will be captured in a binary fashion (i.e. PRESENT or NOT PRESENT) on the CRF by the physician during manual auscultation - i.e. bronchovesicular, crackles. Normal, adventitious and lack of breath sounds will be annotated in a binary fashion (i.e. PRESENT or NOT PRESENT) on the CRF by the independent physician during remote auscultation - i.e. bronchovesicular, crackles

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided